CLINICAL TRIAL: NCT01912989
Title: Motivational Interviewing in NOURISH for Parents of Overweight Children
Acronym: NOURISH+MI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13CRP14570008
Record Dates: First submitted 2013-06-28; First posted 2013-07-31 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Overweight and Obesity
Keywords: motivational interviewing; obesity; parent
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental): NOURISH+ plus motivational interviewing
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: Lifestyle counseling — Parents will participate in one telephone and one in person session of motivational interviewing prior to their participation in an 8 week parent-exclusive treatment focusing on parenting skills to improve their child's overweight.

SUMMARY:
The purpose of this study is to investigate if a brief, motivational interviewing intervention (NOURISH+MI) can improve retention and treatment adherence for parents enrolled in an intervention for their child's overweight (NOURISH+). The investigators hypothesize that children whose parents participate in NOURISH+MI will demonstrate lower attrition and greater adherence with NOURISH+, ultimately leading to greater treatment effects, compared with children whose parents are randomized to NOURISH+ or a control group.

DETAILED DESCRIPTION:
There is an urgent need for innovative approaches to pediatric obesity prevention and treatment. There is also a demand for targeted strategies that reduce attrition and improve compliance with obesity treatment. Intervening exclusively with parents of overweight children is a novel treatment approach, with demonstrated efficacy in reducing child body mass index (BMI) percentile. Motivational interviewing (MI), a brief communication style for exploring and resolving ambivalence about change, may enhance treatment engagement when implemented as part of obesity interventions. Further research investigating MI within pediatric obesity treatments is needed. In the current application, the investigators are examining whether MI implemented with parents for the treatment of their children's overweight can improve treatment effects. NOURISH+, a recently funded R01 (Nourishing Our Understanding of Role modeling to Improve Support and Health; PI, Mazzeo), is a culturally tailored parent intervention for overweight children ages 5-11. NOURISH+ targets lower-income, African American participants, a group at increased risk for pediatric overweight and associated complications, and builds on pilot work which yielded significant reductions in child BMI percentile. The investigators are adding an MI treatment into NOURISH+. Specifically, we will randomly select 60 parents at enrollment and investigate if adding two brief MI sessions prior to the NOURISH+ group intervention will enhance treatment effects. The investigators will be able to compare NOURISH+MI with participants from the two R01 treatment conditions (NOURISH+ and Control), matched on child ethnicity and gender. The investigators hypothesize that children whose parents participate in NOURISH+ MI will demonstrate lower attrition and greater compliance with NOURISH+, ultimately leading to greater treatment effects, compared with children whose parents are randomized to NOURISH+ or a control group.

ELIGIBILITY:
Inclusion Criteria:

* parents/caregivers must be at least 18 years old
* have a child between the ages of 5 and 11
* have a child with a BMI > the 85th%ile
* the eligible child primarily resides in the caregiver's home
* English speaking

Exclusion Criteria:

* non-ambulatory
* pregnant
* have a medical condition that might be negatively impacted by exercise have a psychiatric diagnosis that would impair their ability to respond to assessments or participate in a group
* Parents whose children have a medical or developmental condition that precludes weight loss using conventional diet and exercise methods are also ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of sessions attended | 8 weeks and 4-month follow up

SECONDARY OUTCOMES:
Baseline child dietary intake and change in intake | baseline, 8 weeks, 4 month post
Baseline child physical activity and change in activity | baseline, 8 weeks, 4-month post
Baseline child BMI percentile and change in BMI | baseline, 8 weeks, 4-month post
Baseline parent BMI and change in BMI | baseline, 8 weeks, 4-month post
Baseline parent dietary intake and change in intake | baseline, 8 weeks, 4-month post
Baseline parent physical activity and change in activity | baseline, 8 weeks, 4-month post

CONTACTS AND LOCATIONS:
Overall Officials: Melanie K Bean, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Background] Bean MK, Jeffers AJ, Tully CB, Thornton LM, Mazzeo SE. Motivational interviewing with parents of overweight children: study design and methods for the NOURISH + MI study. Contemp Clin Trials. 2014 Mar;37(2):312-21. doi: 10.1016/j.cct.2014.02.001. Epub 2014 Feb 12. PMID 24530488